CLINICAL TRIAL: NCT02849535
Title: Impact of the PRISM-care Multidisciplinary Oncology Program Versus Usual Care on Secured Drug Intake of Patients With Kidney Cancer, Through Self-management of Adverse Events Related to Oral Targeted Therapies, Control of Drug Interactions, and Sharing of the Information Between Ambulatory and Hospital Settings.
Brief Title: Impact of the PRISM-care Multidisciplinary Oncology Program on Secured Drug Intake of Patients With Kidney Cancer
Acronym: PRISM care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL14_0453
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Oral chemotherapy; Relative dose intensity; Health related program; Secured drug intake
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRISM care program (Experimental): PRISM care is a multidisciplinary program that includes sessions with a hospital pharmacist about the oral chemotherapy: information is given to the patient on adverse events occurrence and management, optimizing drug dosage plan, including drug-drug interactions. Physical sessions will be planned at the beginning of month 1, month 2 and month 3 after the inclusion, then telephone interviews of physical sessions will be planned at month 4, month 5 and month 6. During all these sessions and during the final physical session at the end of month 6, data will be recorded for outcomes assessment.
  Interventions: Behavioral: PRISM care program
- Standard of care (No Intervention): In the group with standard of care, patients will have interviews with a hospital pharmacist only dedicated to the record of data for outcomes assessment. These sessions will be planned at the beginning of month 1, month 2 and month 3 after the inclusion , and at the end at month 6 after the final physical session.

INTERVENTIONS:
Behavioral: PRISM care program — PRISM care is a multidisciplinary program that includes sessions with a hospital pharmacist about the oral chemotherapy: information is given to the patient on adverse events occurrence and management, optimizing drug dosage plan, including drug-drug interactions. Physical sessions will be planned at the beginning of month 1, month 2 and month 3 after the inclusion, then telephone interviews of physical sessions will be planned at month 4, month 5 and month 6. During all these sessions and during the final physical session at the end of month 6, data will be recorded for outcomes assessment.
  Arms: PRISM care program

SUMMARY:
The rise of oral targeted therapies favors outpatient care of cancer patients but exposes them to new risks compared to the injectable chemotherapy in the hospital: non-adherence to treatment, inappropriate management of side effects and interactions with other co-prescribed drugs. The clinical consequences (reduced efficacy and potentialized toxicity) are all the more important that ambulatory monitoring of treatments prescribed at the hospital remains underdeveloped due to default of coordination between these two settings.

Adverse drug reactions are a major concern, as such, and because they involve prescription changes (dose reduction, treatment interruption). This results in a decrease in the dose taken and a risk of loss of efficacy.

In the context of metastatic renal cell carcinoma, the risk of iatrogenicity is even higher because the oral targeted therapies available in this indication have a safety profile marked by potentially serious toxicities (hematologic and cardiac toxicity) or are known to reduce the treatment adherence (digestive and skin toxicities). In addition, these molecules are metabolized by the CYP3A4 hepatic cytochrome, which leads to avoid associating them with drugs inducing and / or inhibiting the CYP3A4, because of the risk of toxicity and / or loss of efficacy.

The investigators propose to assess a program set up to secure drug taking by enhancing self-management of side effects and control of drug interactions by the patient. This program includes pharmaceutical visits and involves inpatient and outpatient (doctor, referent pharmacist and liberal nurse) professionals.

The hypothesis of the study is that the PRISM care program will improve self-management of side effects by the patient, resulting in a relative dose intensity of oral chemotherapy improved compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years old or more
* With metastatic renal cell carcinoma
* With an initiation or change of oral targeted therapy, especially: tyrosine kinase inhibitor (sunitinib, sorafenib, pazopanib, axitinib) or mTor inhibitor (everolimus)
* With ambulatory status (not hospitalized for the management and treatment of its metastatic renal cell carcinoma)
* Without either cognitive disorders or major psychiatric disorders
* With a sufficient autonomy for the management of medication at home
* Having declared an outpatient doctor
* Having declared a usual pharmacy
* Having given his written consent to participate in the study

Exclusion Criteria:

* Significant cognitive and psychiatric disorders
* Management of medication at home exclusively performed by the family caregiver
* Patient in an institution or under guardianship, major protected by law
* Patient refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2017-10-17 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Relative dose intensity of oral chemotherapy | 6 months from the treatment initiation
  Relative dose intensity will be computed by the ratio between the overall dose delivered and the overall dose prescribed during the 6 months of follow-up.

SECONDARY OUTCOMES:
Adherence to the oral chemotherapy measured with the prescription renewal rate | 6 months from the treatment initiation
  Adherence will be measured with the prescription renewal rate by the ambulatory pharmacy (adherence will be defined as a rate ≥80%).
Adherence to the oral chemotherapy measured with the Girerd questionnaire | 6 months from the treatment initiation
  the Girerd questionnaire is a medication adherence questionnaire
Grade 3 and 4 adverse events related to the oral chemotherapy | 6 months from the treatment initiation
Drug interactions (for patients included in the interventional group) | 6 months from the treatment initiation
Cause of changes dose relative intensity: number of reduction of dosage | 6 months from the treatment initiation
Cause of changes dose relative intensity: number of interruption or discontinuation of treatment | 6 months from the treatment initiation
Number of unplanned hospitalizations related to the oral chemotherapy | 6 months from the treatment initiation
Number of emergency admissions related to the oral chemotherapy | 6 months from the treatment initiation
Consumption of health care resources: number and nature of consultations with GPs and / or medical specialists | 6 months from the treatment initiation
Consumption of health care resources: number of acts of biology | 6 months from the treatment initiation
Consumption of health care resources: number of acts of imagery | 6 months from the treatment initiation
Consumption of health care resources: number of prescribed drugs and self-medication and other health products | 6 months from the treatment initiation
Quality of life, measured with the EORTC QLQ-C30 questionnaire (version 3.0) | Inclusion and 6 months from the treatment initiation
Satisfaction with treatment with medicines, measured with the SAT-MED Q questionnaire | Inclusion and 6 months from the treatment initiation
Rate of patients presenting satisfying knowledge about adverse effects of their oral chemotherapy, according to the hospital pharmacists and measured with a 4-items Likert scale | 2 months and 6 months from the treatment initiation
Health locus of control, measured with the Therapeutic Self Care Toll (TSCT) scale | Inclusion and 6 months from the treatment initiation
Patient's perception of its illness, measured with the Brief Illness Perception Questionnaire (B-IPQ) | Inclusion and 6 months from the treatment initiation
Involvement of outpatient caregivers (doctors, pharmacists and liberal nurses) in the PRISM care program | During the 6 months of follow-up
  Involvement will be described by the number and type of: interventions recorded on a dedicated form, solicitations of hospital staff, treatment modifications realized in concertation between oncologist and outpatient doctor.
Satisfaction of outpatient caregivers (doctors, pharmacists and liberal nurses) relative to the PRISM care program, measured with a rating out of 10 | 6 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Catherine RIOUFOL, PharmD PhD, Principal Investigator — Hospices Civils de Lyon
Locations (12):
- France (12):
  - Institut de Cancérologie de l'Ouest, Angers
  - CH de Chambéry, Chambéry
  - Centre de Lutte Contre le Cancer Jean Perrin, Clermont-Ferrand
  - Centre Léon Bérard, Lyon
  - Hôpital Arnaud de Villeneuve, Montpellier
  - APHP Hôpital de la Pitié Salpétrière, Paris
  - Hospices Civils de Lyon Groupement Hospitalier Sud Service pharmaceutique Unité de Pharmacie Clinique Oncologique Pavillon Marcel Bérard 1G 165 chemin du Grand Revoyet, Pierre-Bénite
  - Institut Jean Godinot de Reims, Reims
  - CHU, Rouen
  - ICL Institut de Cancérologie de la Loire Lucien Neuwirth, Saint-Priest-en-Jarez
  - Hôpital Bretonneau, Tours
  - CH Lacari, Vichy